CLINICAL TRIAL: NCT03582865
Title: Genetic Study of CYP2D6 Enzyme and Therapeutic Drug Monitoring of Tamoxifen in Premenopausal Women With Breast Cancer
Brief Title: Genetic Study of CYP2D6 Enzyme and Therapeutic Drug Monitoring of Tamoxifen
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Fawzy Taha, Assistant Lecturer, Assiut University
Other Study IDs: Genetic study and TDM
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Genotyping; Tamoxifen
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- responding: patients who received Tamoxifen 20 mg daily for at least 3 years with good response (no relapse) to tamoxifen. Both genotyping assessment and TDM of tamoxifen and its metabolites will be performed and correlated with the records. Follow up for these patients for further assessment of tamoxifen effectiveness will be carried out for 1- 2 years.
  Interventions: Drug: Tamoxifen 20 mg
- relapse: patients who received Tamoxifen 20 mg daily for at least 3 years who were good responder to the drug but then the response has been diminished (relapse) and they have been shifted to another therapy. They will be exposed to genotyping study of CYP 2D6 to recognize the phenotyping style of that patient that may explain diminishing of response to tamoxifen therapy.
  Interventions: Drug: Tamoxifen 20 mg
- tamoxifen resistant: patients who received Tamoxifen 20 mg daily for not more than 1 year with poor response to tamoxifen (early relapse) and clinically will be shifted to use another medication as they were diagnosed as tamoxifen resistant. Like the second group, they will be exposed to genotyping study of CYP2D6 with the same concept.
  Interventions: Drug: Tamoxifen 20 mg

INTERVENTIONS:
Drug: Tamoxifen 20 mg — Tamoxifen 20 mg is a selective estrogen receptor modulator
  Other Names: Genetic

SUMMARY:
Aim of work:

1. To estimate the frequency of Cyp2D6*1 and *4 alleles in Egyptian patients maintained on tamoxifen (20 mg/day) for management of ER +ve breast cancer.
2. To measure levels of tamoxifen, 4-hydroxy tamoxifen, N-desmethyl-tamoxifen and 4- hydroxyl-N-desmethyl-tamoxifen (endoxifen) in the serum of these patients.
3. To correlate between the levels of tamoxifen/active metabolite enoxifen ratio and CYP2D6*1,*4 genotyping.
4. To investigate which is more valuable investigatory tool for prediction of the clinical outcome (response and/or toxicity) in these patients; either the measurements related to pharmacokinetics: tamoxifen/endoxifen levels or the pharmacogenetic analysis of CYP2D6 *1,*4.

DETAILED DESCRIPTION:
Breast cancer is considered to be the most common cancer among women worldwide. The majority of breast cancer cases (almost 80%) are classified as hormone-dependent cancer, since estrogen, acting via estrogen receptor alpha (ER-α) or estrogen receptor beta (ER-β), is the major inducer of the development and growth of the tumor. These are also called ER-positive breast cancers. The remaining cases are not induced by estrogen and are classified as hormone-independent, or ER-negative, cancers. Since the growth of hormone-dependent cancer cells can be down-regulated by the oppositely active hormones, several endocrine therapies that limit the actions of estrogen (through blocking its production or its receptors) have been developed over the past years. These endocrine therapies have played an important part in treating and improving the outcomes of women with all stages of the disease . Selective estrogen receptor modulators (SERMs) have also been studied for their anti-cancer activity.

Selective estrogen receptor modulators (SERMs) are a class of drugs that act on the estrogen receptor (ER); a characteristic that distinguishes these substances from pure ER agonists and antagonists as their action is different in various tissues, thereby granting the possibility to selectively inhibit or stimulate estrogen-like action in various tissues .

Tamoxifen, which is a SERM, is important for the treatment and prevention of estrogen receptor (ER) positive breast cancer commonly in premenopausal women. It has been shown to decrease disease recurrence and mortality rates by as much as 50% and 30% respectively. It has been also used as a prophylactic treatment for patients who are at high risk of developing breast cancer. Post-menopausal breast cancer patients are commonly treated nowadays with aromatase inhibitors (AIs) for 5 years, alone or combined with tamoxifen for a 3-5 year period. Tamoxifen monotherapy in postmenopausal women with breast cancer may be used for 10 years if the side effects from AIs are too bothersome .

Besides acting as SERMs, it has recently been found that some of tamoxifen's metabolites (as norendoxifen) also act as aromatase inhibitors in vitro. Aromatase converts steroids (e.g., testosterone to estradiol), the inhibition of which severely decreases the amount of available estrogen in the body .

The most common side effects of Tamoxifen:

* Hot flashes, the most common side effect of tamoxifen, affect up to 80% of women.
* Increased risk of endometrial hyperplasia and polyps
* Increased risk for cataract.
* Increased risk for thromboembolic events as well as clinical depression .

Pharmacokinetics of tamoxifen and its clinical implications:

Tamoxifen is a prodrug that is metabolized by several cytochrome P450 enzymes. It is a relatively weak antiestrogen in comparison to its active metabolites, particularly endoxifen. Two parallel pathways bioactivate tamoxifen to endoxifen (4-OH-N-desmethyltamoxifen) through several overlapping cytochrome P450 (CYP) enzymes; primarily CYP3A4/5 and CYP2D6.

For many years, 4-hydroxy-tamoxifen has believed to be primarily responsible for the clinical activity; however, the CYP2D6 metabolites 4-hydroxy-tamoxifen and endoxifen (4-OH-N-desmethyl-tamoxifen) have equal affinity for the estrogen receptor. Because serum concentrations of endoxifen are 6 to 12 times higher than 4-hydroxy-tamoxifen in patients receiving long-term tamoxifen therapy, many think endoxifen is the most significant tamoxifen metabolite.

The rate limiting step in tamoxifen metabolism is catalyzed by the highly polymorphic CYP2D6 enzyme so that CYP2D6 genotype can be translated into predicted metabolic activity phenotypes: poor metabolizer (PM), intermediate metabolizer (IM), extensive metabolizer (EM), ultrarapid metabolizer (UM), which are strongly predictive of endoxifen concentration during tamoxifen treatment.

There is substantial variation in CYP2D6 genotypes among different populations. CYP2D6*1 is the wild-type allele and is associated with normal enzyme activity and the normal "extensive metabolizer" phenotype. The CYP2D6 alleles *2, *33, and *35 are also considered to have near-normal activity. Other alleles include variants that produce a non-functioning enzyme (e.g., *3, *4, *5, and *6) or an enzyme with reduced activity (e.g., *10, *17, and *41). There are large inter-ethnic differences in the frequency of these alleles, with *3, *4, *5, *6, and *41 being more common in the Caucasian population, *17 more common in Africans, and *10 more common in Asians. Also it was found that *1 and *4 alleles are more common in Egyptians.

Patients with low-activity CYP2D6 phenotypes have substantially lower endoxifen steady-state concentrations . It is unclear whether patients with genotypes that confer low CYP2D6 activity have inferior efficacy from tamoxifen treatment, but if so, preemptive genotyping to guide tamoxifen dose selection could be a viable strategy to improve treatment effectiveness.

Despite the proven efficacy of tamoxifen, some women experience cancer recurrence during or after treatment. Therapeutic failure may be caused by tumor resistance to antiestrogen therapy or inadequate bioactivation of tamoxifen to its active metabolite, endoxifen.

Some studies have reported that patients with low endoxifen concentrations (below 5.9 ng/ml) have increased the risk of inferior tamoxifen efficacy with consequent cancer recurrence compared with its concentration in intermediate and rapid or ultra-rapid metabolizers taking the same dose. This can open the way for application of therapeutic drug monitoring of tamoxifen and its metabolite endoxifen for possible dose escalation especially a fixed dose of the drug is usually used which is 20 mg/day.

The issue of relying on genotyping profile of CYP2D6 and its variants or use of TDM of tamoxifen and its metabolite endoxifen or the combination of both parameters to correlate with clinical response, adverse effect and dose modification of tamoxifen is still under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal patients will be included in this study, with hormone receptor positive tumors.
* The hormone receptor positive tumor is diagnosed by microscopic examination if ≥ 10% of the cells are positive for estrogen by immunohistochemistry analysis.
* All patients with normal hepatic and renal function, aspartate aminotransferase and alanine aminotransferase (≤2 upper normal limit) and serum creatinine (≤1.2 mg/dl).

Exclusion Criteria:

* Patients treated with other hormonal therapy, radiation or chemotherapy will be excluded from the study.
* Pregnant or breast feeding women will be excluded from the study.
* Patients who are taking drugs that are known to inhibit CYP2D6 activity as SSRIs will be excluded from the study.

Ages: 20 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Premenopausal women suffering from breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Estimate the frequency of Cyp2D6*1 and *4 alleles in Egyptian patients maintained on tamoxifen (20 mg/day) for management of ER +ve breast cancer. | 6 months
  The CYP2D6 genotypes will be determined using the TaqMan Allelic Discrimination Assay.

SECONDARY OUTCOMES:
measuring levels of tamoxifen, 4-hydroxy tamoxifen, N-desmethyl-tamoxifen and 4- hydroxyl-N-desmethyl-tamoxifen (endoxifen) in the serum ofbreast cancer patients. | 2 months
  Plasma concentrations of tamoxifen, 4-hydroxy-tamoxifen (4-OH-tam), N-desmethyl-tamoxifen (N-DM-tam) and 4-hydroxy-N-desmethyl-tamoxifen (endoxifen) will be measured using sensitive HPLC-PDA assay method.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Taha, Principal Investigator — Assiut University; Ehab Eldesoky, Study Director — Assiut University; Mohammad Hareedy, Study Director — Assiut University

REFERENCES:
- [Background] Johnston SR. New strategies in estrogen receptor-positive breast cancer. Clin Cancer Res. 2010 Apr 1;16(7):1979-87. doi: 10.1158/1078-0432.CCR-09-1823. Epub 2010 Mar 23. PMID 20332324
- [Background] Davies C, Pan H, Godwin J, Gray R, Arriagada R, Raina V, Abraham M, Medeiros Alencar VH, Badran A, Bonfill X, Bradbury J, Clarke M, Collins R, Davis SR, Delmestri A, Forbes JF, Haddad P, Hou MF, Inbar M, Khaled H, Kielanowska J, Kwan WH, Mathew BS, Mittra I, Muller B, Nicolucci A, Peralta O, Pernas F, Petruzelka L, Pienkowski T, Radhika R, Rajan B, Rubach MT, Tort S, Urrutia G, Valentini M, Wang Y, Peto R; Adjuvant Tamoxifen: Longer Against Shorter (ATLAS) Collaborative Group. Long-term effects of continuing adjuvant tamoxifen to 10 years versus stopping at 5 years after diagnosis of oestrogen receptor-positive breast cancer: ATLAS, a randomised trial. Lancet. 2013 Mar 9;381(9869):805-16. doi: 10.1016/S0140-6736(12)61963-1. PMID 23219286
- [Background] Dowsett M, Cuzick J, Ingle J, Coates A, Forbes J, Bliss J, Buyse M, Baum M, Buzdar A, Colleoni M, Coombes C, Snowdon C, Gnant M, Jakesz R, Kaufmann M, Boccardo F, Godwin J, Davies C, Peto R. Meta-analysis of breast cancer outcomes in adjuvant trials of aromatase inhibitors versus tamoxifen. J Clin Oncol. 2010 Jan 20;28(3):509-18. doi: 10.1200/JCO.2009.23.1274. Epub 2009 Nov 30. PMID 19949017
- [Background] Goldhirsch A, Winer EP, Coates AS, Gelber RD, Piccart-Gebhart M, Thurlimann B, Senn HJ; Panel members. Personalizing the treatment of women with early breast cancer: highlights of the St Gallen International Expert Consensus on the Primary Therapy of Early Breast Cancer 2013. Ann Oncol. 2013 Sep;24(9):2206-23. doi: 10.1093/annonc/mdt303. Epub 2013 Aug 4. PMID 23917950
- [Background] Lu WJ, Xu C, Pei Z, Mayhoub AS, Cushman M, Flockhart DA. The tamoxifen metabolite norendoxifen is a potent and selective inhibitor of aromatase (CYP19) and a potential lead compound for novel therapeutic agents. Breast Cancer Res Treat. 2012 May;133(1):99-109. doi: 10.1007/s10549-011-1699-4. Epub 2011 Aug 4. PMID 21814747
- [Background] Klein DJ, Thorn CF, Desta Z, Flockhart DA, Altman RB, Klein TE. PharmGKB summary: tamoxifen pathway, pharmacokinetics. Pharmacogenet Genomics. 2013 Nov;23(11):643-7. doi: 10.1097/FPC.0b013e3283656bc1. No abstract available. PMID 23962908
- [Background] Johnson MD, Zuo H, Lee KH, Trebley JP, Rae JM, Weatherman RV, Desta Z, Flockhart DA, Skaar TC. Pharmacological characterization of 4-hydroxy-N-desmethyl tamoxifen, a novel active metabolite of tamoxifen. Breast Cancer Res Treat. 2004 May;85(2):151-9. doi: 10.1023/B:BREA.0000025406.31193.e8. PMID 15111773
- [Background] Murdter TE, Schroth W, Bacchus-Gerybadze L, Winter S, Heinkele G, Simon W, Fasching PA, Fehm T; German Tamoxifen and AI Clinicians Group; Eichelbaum M, Schwab M, Brauch H. Activity levels of tamoxifen metabolites at the estrogen receptor and the impact of genetic polymorphisms of phase I and II enzymes on their concentration levels in plasma. Clin Pharmacol Ther. 2011 May;89(5):708-17. doi: 10.1038/clpt.2011.27. Epub 2011 Mar 30. PMID 21451508
- [Background] Gaedigk A, Simon SD, Pearce RE, Bradford LD, Kennedy MJ, Leeder JS. The CYP2D6 activity score: translating genotype information into a qualitative measure of phenotype. Clin Pharmacol Ther. 2008 Feb;83(2):234-42. doi: 10.1038/sj.clpt.6100406. Epub 2007 Oct 31. PMID 17971818
- [Background] Borges S, Desta Z, Jin Y, Faouzi A, Robarge JD, Philips S, Nguyen A, Stearns V, Hayes D, Rae JM, Skaar TC, Flockhart DA, Li L. Composite functional genetic and comedication CYP2D6 activity score in predicting tamoxifen drug exposure among breast cancer patients. J Clin Pharmacol. 2010 Apr;50(4):450-8. doi: 10.1177/0091270009359182. Epub 2010 Jan 15. PMID 20081063
- [Background] Saladores P, Murdter T, Eccles D, Chowbay B, Zgheib NK, Winter S, Ganchev B, Eccles B, Gerty S, Tfayli A, Lim JS, Yap YS, Ng RC, Wong NS, Dent R, Habbal MZ, Schaeffeler E, Eichelbaum M, Schroth W, Schwab M, Brauch H. Tamoxifen metabolism predicts drug concentrations and outcome in premenopausal patients with early breast cancer. Pharmacogenomics J. 2015 Feb;15(1):84-94. doi: 10.1038/tpj.2014.34. Epub 2014 Aug 5. PMID 25091503
- [Background] Hertz DL, Snavely AC, McLeod HL, Walko CM, Ibrahim JG, Anderson S, Weck KE, Magrinat G, Olajide O, Moore S, Raab R, Carrizosa DR, Corso S, Schwartz G, Peppercorn JM, Evans JP, Jones DR, Desta Z, Flockhart DA, Carey LA, Irvin WJ Jr. In vivo assessment of the metabolic activity of CYP2D6 diplotypes and alleles. Br J Clin Pharmacol. 2015 Nov;80(5):1122-30. doi: 10.1111/bcp.12665. Epub 2015 Aug 2. PMID 25907378
- [Background] de Vries Schultink AH, Zwart W, Linn SC, Beijnen JH, Huitema AD. Effects of Pharmacogenetics on the Pharmacokinetics and Pharmacodynamics of Tamoxifen. Clin Pharmacokinet. 2015 Aug;54(8):797-810. doi: 10.1007/s40262-015-0273-3. PMID 25940823
- [Background] Goetz MP, Suman VJ, Hoskin TL, Gnant M, Filipits M, Safgren SL, Kuffel M, Jakesz R, Rudas M, Greil R, Dietze O, Lang A, Offner F, Reynolds CA, Weinshilboum RM, Ames MM, Ingle JN. CYP2D6 metabolism and patient outcome in the Austrian Breast and Colorectal Cancer Study Group trial (ABCSG) 8. Clin Cancer Res. 2013 Jan 15;19(2):500-7. doi: 10.1158/1078-0432.CCR-12-2153. Epub 2012 Dec 4. PMID 23213055
- [Background] Schroth W, Goetz MP, Hamann U, Fasching PA, Schmidt M, Winter S, Fritz P, Simon W, Suman VJ, Ames MM, Safgren SL, Kuffel MJ, Ulmer HU, Bolander J, Strick R, Beckmann MW, Koelbl H, Weinshilboum RM, Ingle JN, Eichelbaum M, Schwab M, Brauch H. Association between CYP2D6 polymorphisms and outcomes among women with early stage breast cancer treated with tamoxifen. JAMA. 2009 Oct 7;302(13):1429-36. doi: 10.1001/jama.2009.1420. PMID 19809024
- [Background] Nakamura Y, Ratain MJ, Cox NJ, McLeod HL, Kroetz DL, Flockhart DA. Re: CYP2D6 genotype and tamoxifen response in postmenopausal women with endocrine-responsive breast cancer: the Breast International Group 1-98 trial. J Natl Cancer Inst. 2012 Aug 22;104(16):1264; author reply 1266-8. doi: 10.1093/jnci/djs304. Epub 2012 Jul 31. No abstract available. PMID 22851270
- [Background] Robinson DR, Wu YM, Vats P, Su F, Lonigro RJ, Cao X, Kalyana-Sundaram S, Wang R, Ning Y, Hodges L, Gursky A, Siddiqui J, Tomlins SA, Roychowdhury S, Pienta KJ, Kim SY, Roberts JS, Rae JM, Van Poznak CH, Hayes DF, Chugh R, Kunju LP, Talpaz M, Schott AF, Chinnaiyan AM. Activating ESR1 mutations in hormone-resistant metastatic breast cancer. Nat Genet. 2013 Dec;45(12):1446-51. doi: 10.1038/ng.2823. Epub 2013 Nov 3. PMID 24185510
- [Background] Li S, Shen D, Shao J, Crowder R, Liu W, Prat A, He X, Liu S, Hoog J, Lu C, Ding L, Griffith OL, Miller C, Larson D, Fulton RS, Harrison M, Mooney T, McMichael JF, Luo J, Tao Y, Goncalves R, Schlosberg C, Hiken JF, Saied L, Sanchez C, Giuntoli T, Bumb C, Cooper C, Kitchens RT, Lin A, Phommaly C, Davies SR, Zhang J, Kavuri MS, McEachern D, Dong YY, Ma C, Pluard T, Naughton M, Bose R, Suresh R, McDowell R, Michel L, Aft R, Gillanders W, DeSchryver K, Wilson RK, Wang S, Mills GB, Gonzalez-Angulo A, Edwards JR, Maher C, Perou CM, Mardis ER, Ellis MJ. Endocrine-therapy-resistant ESR1 variants revealed by genomic characterization of breast-cancer-derived xenografts. Cell Rep. 2013 Sep 26;4(6):1116-30. doi: 10.1016/j.celrep.2013.08.022. Epub 2013 Sep 19. PMID 24055055
- [Background] Lien EA, Ueland PM, Lonning PE. Re: Active tamoxifen metabolite plasma concentrations after coadministration of tamoxifen and the selective serotonin reuptake inhibitor paroxetine. J Natl Cancer Inst. 2004 Jun 2;96(11):884; author reply 884-5. doi: 10.1093/jnci/djh160. No abstract available. PMID 15173277
- [Background] Lim YC, Desta Z, Flockhart DA, Skaar TC. Endoxifen (4-hydroxy-N-desmethyl-tamoxifen) has anti-estrogenic effects in breast cancer cells with potency similar to 4-hydroxy-tamoxifen. Cancer Chemother Pharmacol. 2005 May;55(5):471-8. doi: 10.1007/s00280-004-0926-7. Epub 2005 Feb 1. PMID 15685451